CLINICAL TRIAL: NCT02003716
Title: Use of the DeFRA Questionnaire as a "Primary Anamnestic Form" Through a Large Scale Screening of the Population
Brief Title: DeFRA Questionnaire as an Anamnestic Form
Status: Completed | Type: Observational
Sponsor: Valmontone Hospital (Other)
Responsible Party: Principal Investigator, Dell'anna Vincenzo, Principal Investigator, Valmontone Hospital
Other Study IDs: VDA-001-2012
Record Dates: First submitted 2013-11-19; First posted 2013-12-06 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The DeFRA questionnaire is a new validated algorithm derived from FRAX. Here we use the DeFRA as a "primary anamnestic from" to identify subjects at risk of osteoporosis in a population never screened before and never treated for this disease.

DETAILED DESCRIPTION:
There is an increasing recognition that the management of osteoporosis requires the characterization of fracture risk to be based on absolute risk rather than single measures such as bone mineral density (BMD). However, the threshold for pharmacological intervention for osteoporosis remains controversial.

The aim of the present project is to perform a large scale study to identify subjects at risk of osteoporosis by administering the DeFRA questionnaire in a population never screened or treated before for osteoporosis.

DeFRA questionnaire will be administered before and after DEXA scanning, to further validate the questionnaire and to highlight the predictive value of this protocol as a tool to screen the general population.

ELIGIBILITY:
Inclusion Criteria:

* age: 50 to 70 years
* no overt pathologies
* never screened before for osteoporosis
* no prior use of drugs for osteoporosis
* signed informed consent form

Exclusion Criteria:

* overt pathologies (cancer, neurodegenerative diseases, renal or hepatic insufficiency)
* use of the following drugs: cortisones, loop diuretics, antiepileptic drugs, aromatase inhibitors, dicoumarols, thyroxin in suppressive therapy, antiosteoporosis drugs)
* patients who underwent radiation therapy
* hypercalcemia or alterations of the phospho-calcic metabolism
* patients with metabolic diseases of the bone (including hyperparathyroidism or Paget disease)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general population, never screened before for osteoporosis and never subject to treatment
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
percent risk of a fracture | day 1
  The DeFRA questionnaire is administered within the same day with or without the DeXA measurement, to evaluate statistically significant differences in the percent risk of a fracture

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Dell'Anna, Dr., Principal Investigator — Valmontone Hospital
Locations (1):
- Valmontone Hospital, Valmontone, Roma, Italy